CLINICAL TRIAL: NCT00931957
Title: Etanercept: Single Blind Control Study in Ocular Manifestations of Behcet's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Fereydoun Davatchi, Head Rheumatology Research Center, Rheumatology Research Center, Tehran University for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 860241-5807
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Behcet Syndrome; Uveal Disease
Keywords: Etanercept; Behcet's syndrome; Behcet's Disease; Ocular Lesions; Uveitis; Retinal Vasculitis
MeSH Terms: conditions — Behcet Syndrome; Uveal Diseases; Uveitis; Retinal Vasculitis | interventions — Etanercept; Methotrexate; Prednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept-MTX-Prednisolone (Active Comparator): Methotrexate + Prednisolone + Etanercept
  Interventions: Drug: Etanercept, Methotrexate, Prednisolone
- B, MTX-Prednisolone (Other): Methotrexate + Prednisolone
  Interventions: Drug: Etanercept, Methotrexate, Prednisolone

INTERVENTIONS:
Drug: Etanercept, Methotrexate, Prednisolone — In: Arm A, Etanercept-MTX-Prednisolone:
  Etanercept 50 mg weekly (subcutaneous injection) for 12 months. Methotrexate 15 mg weekly for 12 months. Prednisolone: 30 mg daily, in divided doses, as initial dose. The dose will be reduced and adjusted to the eye's inflammation. Discontinuation if no inflammation with very low doses.
  In Arm B:
  Methotrexate 15 mg weekly for 12 months. Prednisolone: 30 mg daily, in divided doses, as initial dose. The dose will be reduced and adjusted to the eye's inflammation. Discontinuation if no inflammation with very low doses.
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to find if Etanercept can improve the outcome of ocular lesions of Behcet's Disease treated with Methotrexate and Prednisolone

DETAILED DESCRIPTION:
To test in a randomized single blind control trial the efficacy of Etanercept in patients with posterior uveitis and/or retinal vasculitis of Behcet's disease treated with Methotrexate and prednisolone

ELIGIBILITY:
Inclusion Criteria:

* Behcet's Disease according to the International Criteria for Behcet's disease (ICBD)
* Active posterior uveitis and/or retinal vasculitis

Exclusion Criteria:

* Visual acuity inferior to 1/10 on Snellen chart
* Being under cytotoxic drugs or having received them in the past 2 months
* Not being able to follow the one year treatment and the regular follow ups

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity, Disease Activity Index (DAI) for Posterior Uveitis, DAI for Retinal vasculitis | One Year

SECONDARY OUTCOMES:
DAI for Anterior Uveitis, Total Inflammatory Acitivity Index, Total Adjusted Disease Activity Index | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, MD, Study Chair — Rheumatology Research Center, Medical Sciences/University of Teheran
Locations (1):
- Rheumatology Research Center, Behcet's Disease Unit (Shariati Hospital), Tehran, Iran

REFERENCES:
- [Background] Melikoglu M, Ozvazgan y Fresko I et al. The response of treatment resistant uveitis in Behcet's syndrome (BS) to a TNF-α blocker, Etanercept: an open study. Arthritis Rheum 2002; 46: S181, (Abstract) 400
- [Background] Davatchi F, Shahram F, Chams H, Jamshidi AR, Nadji A, Chams C, Akbarian M, Gharibdoost F. High dose methotrexate for ocular lesions of Behcet's disease. Preliminary short-term results. Adv Exp Med Biol. 2003;528:579-84. doi: 10.1007/0-306-48382-3_118. No abstract available. PMID 12918769
- [Background] Davatchi F. New and innovative therapies for Behcet's Disease. APLAR Journal of Rheumatology 2004; 7: 141-145
- [Background] Davatchi F, Shams H, Nadji A, Jamshidi AR, Akhlaghi M, Sadeghi Abdollahi B, Ziaie N, Akbarian M, Gharibdoost F. Management of ocular manifestations of Behcet's Disease: outcome with cytotoxic drugs. APLAR Journal of Rheumatology 2005; 8: 119-123
- See also: Rheumatology Research Center, Medical Sciences/University of Tehran — http://rrc.tums.ac.ir/